CLINICAL TRIAL: NCT04596787
Title: The Performance Properties and Efficacy of Ultrasound-Guided Bilateral Thoracic Paravertebral Blocks in Obese and Non-obese Patients Undergoing Reduction Mammaplasty: A Historical Cohort Study
Brief Title: Bilateral Thoracic Paravertebral Blocks in Obese and Non-obese Patients Undergoing Reduction Mammaplasty
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emine Aysu Salviz, MD, MD, Attending Anesthesiologist, Associate Professor, Istanbul University
Other Study IDs: 2020/964
Record Dates: First submitted 2020-10-18; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Pain, Postoperative; Obesity; Thoracic Paravertebral Blocks; Ultrasound; Performance
Keywords: Obesity; Thoracic paravertebral blocks; Ultrasound-guidance; Performance difficulty; Satisfaction
MeSH Terms: conditions — Pain, Postoperative; Obesity; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Obese Patients (Group NO: body mass index (BMI) <30): Patients received bilateral single injection ultrasound (US)-guided bilateral thoracic paravertebral block (TPVB) at the level of T3-T4 with 20 mL bupivacaine 0.375% per injection/side.
  Interventions: Procedure: Bilateral Thoracic paravertebral block
- Obese Patients (Group O: body mass index (BMI) ≥30): Patients received bilateral single injection ultrasound (US)-guided bilateral thoracic paravertebral block (TPVB) at the level of T3-T4 with 20 mL bupivacaine 0.375% per injection/side.
  Interventions: Procedure: Bilateral Thoracic paravertebral block

INTERVENTIONS:
Procedure: Bilateral Thoracic paravertebral block — The blocks were performed at the T3-T4 level bilaterally to block the dermatomes between the T2 and T6 levels (breast innervation area).
  Other Names: TPVBs

SUMMARY:
Aim: Although regional anesthesia (RA) techniques are advantageous in the anesthetic management of obese patients (body mass index (BMI)≥30); their performances can still be associated with technical difficulties and greater failure rates. The aim of this study is to compare the performance properties and analgesic efficacy of ultrasound (US)-guided bilateral thoracic paravertebral blocks (TPVBs) in obese and non-obese patients.

Material methods: After obtaining ethics committee approval; data of 82 patients, who underwent elective bilateral reduction mammaplasty under general anesthesia with adjunctive TPVB analgesia between December of 2016 and February of 2020, were reviewed. Patients were allocated into two groups with respect to their BMI scores (Group NO: BMI<30 and Group O: BMI≥30). Demographics, TPVB ideal US image visualization and performance times, needle tip visualisation and TPVB performance difficulties, number of needle maneuvers, surgical, anesthetic and analgesic follow-up parameters, incidence of postoperative nausea vomiting (PONV), sleep duration, length of postanesthesia care unit (PACU) and hospital stay, patient and surgeon satisfaction scores were all investigated and compared.

DETAILED DESCRIPTION:
Aim: The number of obese patients (body mass index (BMI)≥30) has increased dramatically worldwide, and we, as anesthesiologists, routinely come up against them in our daily clinical practice. Although the preference of various peripheral and neuroaxial regional anesthesia (RA) techniques seems to be advantageous in the anesthetic management of these patients, their performances can also be associated with technical difficulties and greater failure rates. The aim of this study is to compare the performance properties and analgesic efficacy of ultrasound (US)-guided thoracic paravertebral blocks (TPVBs) in obese and non-obese patients.

Material methods: After obtaining ethics committee approval; data of 82 patients, who underwent elective bilateral reduction mammaplasty under general anesthesia with adjunctive TPVB analgesia between December of 2016 and February of 2020, were reviewed. Patients were allocated into two groups with respect to their BMI scores (Group NO: BMI<30 and Group O: BMI≥30). Demographics, TPVB ideal US image visualization and performance times, needle tip visualisation and TPVB performance difficulties, number of needle maneuvers, surgical, anesthetic and analgesic follow-up parameters, incidence of postoperative nausea vomiting (PONV), sleep duration, length of postanesthesia care unit (PACU) and hospital stay, patient and surgeon satisfaction scores were all investigated and compared. Student's t, Mann-Whitney-U and Chi-square tests were used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status of 1-3
* Capable of consenting
* Capable of understanding the instructions for using the NRS pain scores
* Capable of replying the questions
* Lack of contraindications to regional anesthesia (allergy to a LA, local infection, and coagulopathy) and especially TPVB
* Absence of mental/psychiatric disorders
* Absence of chronic analgesic/opioid use
* Absence of alcohol/illicit drug use

Exclusion Criteria:

* Patient refusal of RA/TPVB performance
* American Society of Anesthesiologists (ASA) physical status of 4
* Not capable of consenting
* Not capable of understanding the instructions for using the NRS pain scores
* Not capable of replying the questions
* Contraindications to regional anesthesia (allergy to a LA, local infection, and coagulopathy) and especially TPVB
* Presence of mental/psychiatric disorders
* Presence of chronic analgesic/opioid use
* Presence of alcohol/illicit drug use

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (obese and non-obese) required reduction mammoplasty surgery and received general anesthesia with TPVB analgesia
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Thoracic paravertebral block (TPVB) performance time | 0-20 minutes
  Time period between the US probe placement to the right side at T3-T4 level and the needle withdrawal from the left side T3-T4 level

SECONDARY OUTCOMES:
Postoperative numeric rating scale (NRS) pain scores | 0-24 hours
  NRS pain scores (0: no pain, 10: worst pain imaginable) through postoperative first 24 hours
Ideal US image visualization time | 0-5 minutes
  Time period between the US probe placement at T3-T4 level and visualizing the ideal image to perform the block
Difficulty of needle tip visualization | 0-20 minutes
  Likert scale: 1-5 (1:very poor, 5:very good)
Number of needle maneuvers to reach the paravertebral space | 0-20 minutes
  Number of needle maneuvers to reach the paravertebral space (PVS)
Requirement of additional maneuver due to insufficient local anesthetic spread | 0-20 minutes
  Requirement of additional needle maneuver due to insufficient local anesthetic (LA) spread
Difficulty of TPVB according to the anesthesiologists | 0-20 minutes
  Likert scale: 1-5 (1:very poor, 5:very good)
Length of stay in postoanesthesia care unit (PACU) | 0-1 hours
  Modified Aldrete Scoring system (≥9/10)
Number of patients required fentanyl intraoperatively | Intraoperative 2-6 hours
  If a ≥ 20% increase above preinduction values in MAP or HR was observed during the perioperative period, additional fentanyl dose (1 μg/kg) was applied intravenously.
Time to postoperative first pain | 0-48 hours
  Postoperative first pain description (NRS ≥4) until discharge
Number of paracetamol requirement through the postoperative first 24 hours | 0-24 hours
  Paracetamol was used when postoperative pain NRS ≥4 in the postanesthesia care unit or on the wards (on postoperative day 1)
Number of tramadol requirement through the postoperative first 24 hours | 0-24 hours
  Tramadol was used when postoperative pain NRS ≥4 again after 1 hour of paracetamol application in the postanesthesia care unit or on the wards (on postoperative day 1)
Incidence of PONV through the postoperative first 24 hours | 0-24 hours
  Number of feeling nausea or vomiting
Duration of sleep through the postoperative first 24 hours | 0-24 hours
  Total hours of sleep at first night
Length of hospital stay | 0-48 hours
  Post Anaesthetic Discharge Scoring System (PADSS) (≥9/10)
Patient satisfaction | 0-48 hours
  Satisfaction score during hospital discharge: 0: very unsatisfied, 3: very satisfied
Surgeon satisfaction | 0-48 hours
  Satisfaction score during hospital discharge: 0: very unsatisfied, 3: very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Emine A Salviz, Assoc Prof, Principal Investigator — Study Principal Investigator

REFERENCES:
- [Result] Kilicaslan A, Topal A, Erol A, Borazan H, Bilge O, Otelcioglu S. Ultrasound-guided multiple peripheral nerve blocks in a superobese patient. Case Rep Anesthesiol. 2014;2014:896914. doi: 10.1155/2014/896914. Epub 2014 Jan 22. PMID 24587923
- [Result] Franco CD, Gloss FJ, Voronov G, Tyler SG, Stojiljkovic LS. Supraclavicular block in the obese population: an analysis of 2020 blocks. Anesth Analg. 2006 Apr;102(4):1252-4. doi: 10.1213/01.ane.0000198341.53062.a2. PMID 16551933
- [Result] Kula AO, Riess ML, Ellinas EH. Increasing body mass index predicts increasing difficulty, failure rate, and time to discovery of failure of epidural anesthesia in laboring patients. J Clin Anesth. 2017 Feb;37:154-158. doi: 10.1016/j.jclinane.2016.11.010. Epub 2017 Jan 10. PMID 28235511
- [Derived] Salviz EA, Bingul ES, Guzel M, Savran Karadeniz M, Turhan O, Emre Demirel E, Saka E. Comparison of Performance Characteristics and Efficacy of Bilateral Thoracic Paravertebral Blocks in Obese and Non-Obese Patients Undergoing Reduction Mammaplasty Surgery: A Historical Cohort Study. Aesthetic Plast Surg. 2023 Aug;47(4):1343-1352. doi: 10.1007/s00266-023-03270-w. Epub 2023 Feb 10. PMID 36763114